CLINICAL TRIAL: NCT04692038
Title: A Real-World Study to Evaluate the Diagnostic Value of Puncture Biopsy for Peripheral Lung Nodules Under the Guidance of Augmented Reality Navigation System Combined With Radial EBUS
Brief Title: Evaluate the Diagnostic Value of Puncture Biopsy for PPL Under the Guidance of Navigation and Radial EBUS: a Real-World Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Professor, Guangzhou Institute of Respiratory Disease
Other Study IDs: 20201215
Record Dates: First submitted 2020-12-29; First posted 2020-12-31 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Lung; Nodes
Keywords: Peripheral pulmonary nodules; biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment Group: The subjects would receive forceps biopsy combined with puncture biopsy under the guidance of Augmented Reality Navigation and Radial EBUS
  Interventions: Device: Forceps biopsy combined with puncture biopsy under the guidance of Augmented Reality Navigation and Radial EBUS

INTERVENTIONS:
Device: Forceps biopsy combined with puncture biopsy under the guidance of Augmented Reality Navigation and Radial EBUS — During the operation, under the guidance of Augmented Reality Navigation, the bronchoscope will reach the location of the target pulmonary nodules, and the EBUS probe will be inserted through the bronchoscope working channel, and gradually approach the target nodules to obtain EBUS images. After typical EBUS images are observed and the location is confirmed, the EBUS probe will be withdrawn and biopsy forceps and puncture biopsy needle will be used to obtain samples at the target locations respectively.

SUMMARY:
The study is designed to evaluate the safety and effectiveness of biopsy forceps combined with puncture biopsy for the diagnosis of peripheral pulmonary nodules under the guidance of Augmented Reality Navigation System combined with radial endobronchial ultrasound (r-EBUS), and to explore the factors influencing the diagnosis rate.

DETAILED DESCRIPTION:
The study will last for no longer than 12 months. Patients will be first screened, and only after meeting all the inclusion criteria, not meeting any exclusion criteria, and signing the informed consent, could they be enrolled in the group to receive forceps biopsy combined with puncture biopsy to sample the target nodules. The primary endpoint is the combined diagnostic yield of forceps biopsy and puncture biopsy. The secondary endpoints include the success rate of biopsy, the operation time of the bronchoscope and so on.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old; 2. Chest CT shows that the peripheral lung noduleswith uncertain diagnosis are adjacent or far from the airway, and/or are difficult to obtain samples by routine biopsy as assessed by investigators; 3. Understand the research and sign the informed consent form.

Exclusion Criteria:

* 1. Contraindications for bronchoscopy; 2. Severe cardiopulmonary dysfunction and other diseases that may significantly increase the risk of surgery; 3. Bronchoscopy shows visible intra-airway nodules above the 3rd bronchus; 4. The investigator believes that the patient has other conditions that are not suitable for inclusion in this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who meet all inclusion criteria and do not meet any exclusion criteria will be enrolled in the study consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-10 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
Combined Diagnostic yield | Six months
  Diagnostic yield is defined as the proportion of nodules diagnosed by combined technologies in all nodulesundergoing bronchoscopy biopsy.

SECONDARY OUTCOMES:
Diagnostic yield | Six months
  Diagnostic yield is defined as the proportion of nodulesdiagnosed by forceps biopsy (or puncture biopsy) in all nodulesundergoing bronchoscopy biopsy.
The success rate of biopsy | Immediately after bronchoscopy biopsy
  The success rate of biopsy is defined as the number of nodules with at least one qualified abnormal lung tissue that can be used for pathological diagnosis divided by the number of all nodules diagnosed by combined technologies.
Operation time of the bronchoscopy | Immediately after bronchoscopy biopsy
  The operation time of the bronchoscopy is defined as the total time from insertion of the bronchoscope to withdrawal of the bronchoscope.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China